CLINICAL TRIAL: NCT00173524
Title: PharmacoEconomic Assessment IRESSA® in the Treatment of Non-Small-Cell Lung Cancer (NSCLC) : A Cost-Effectiveness Analysis and Cost-Utility Analysis
Brief Title: PharmacoEconomic Assessment IRESSA® in the Treatment of Non-Small-Cell Lung Cancer (NSCLC)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chih-Hsin Yang, National Taiwan University Hospital
Other Study IDs: 9461700718
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFR Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: PharmacoEconomic Assessment — Collecting PE data.

SUMMARY:
The objective of this pharmacoeconomics (PE) study is to evaluate the cost- effectiveness analysis and cost-utility analysis of IRESSA® as first line treatment of NSCLC from the society perspective, based on resources and outcomes from patients who met the inclusion criteria for this naturalistic study comparing to existing first line platinum-based regimen chemotherapy.

DETAILED DESCRIPTION:
Patients with late-stage NSCLC are often symptomatic, with specific pulmonary problems (eg, cough, breathlessness, hemoptysis) and general symptoms (eg. fatigue, weight loss) that can cause extreme distress to the patient. Therefore, improvements in disease-related symptoms and quality of life (QoL) are the key desired outcomes of medical management.7 Effective, palliative, low-toxicity with reasonable treatment cost for patients with advanced NSCLC are needed. Recently, more and more countries consider evidence of economic value along with clinical efficacy.

The epidermal growth factor receptor (EGFR) is a promising target for anticancer therapy because it is expressed or highly expressed in a variety of tumors, including NSCLC. 8,9 Furthermore, high levels of EGFR expression have been associated with a poor prognosis in lung cancer patients in several studies. 10-12 EGFR-targeted cancer therapies are currently being developed; strategies include inhibition of the intracellular tyrosine kinase domain of the receptor by small molecules such as gefitinib (Iressa [ZD1839]; AstraZeneca, Wilmington, DE).13 Iressa is an orally active, selective EGFR tyrosine kinase inhibitor that blocks signal transduction pathways implicated in the proliferation and survival of cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB/IV NSCLC No immediate need for palliative radiotherapy and No prior chemotherapy ; age > 20 Y/O; ECOG PS: 0 - 2; ANC >2000 ; PLT >100k ; Hb > 10; total bilirubin < 2.0 mg/dL; serum creatinine < 2 mg/dl; SGPT and SGOT < 2.5 ×ULN, alkaline phosphatase < 5 ×ULN ; life expectancy >6mos

Exclusion Criteria:

* If the patients have brain metastases or receive radiotherapy, the disease must be stable for more than 6 weeks after the last dose of radiotherapy;
* 2nd malignancies;
* Unable to swallow tablets;
* Patients (M/F) with reproductive potential not implementing adequate contraceptive measurements;
* Pregnant or lactating patients;
* Participation in other clinical trials within 30 days of study entry;
* Major systemic disease which in the investigator's opinion might confound the clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients accrued to a gefitinib first line prospective study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-09; Study Completion 2005-09 (Estimated)

PRIMARY OUTCOMES:
The objective of this PE study is to evaluate the cost- effectiveness analysis and cost-utility analysis of IRESSA® as first line treatment of NSCLC from the society perspective, comparing to existing first line platinum-based regimen chemotherapy. | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zone-Zhe, M.D., Principal Investigator — Department of Oncology , National Taiwan University Hospital; Cheng Ann-Lii, M.D.,Ph.D., Study Chair — Department of Oncology , National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan